CLINICAL TRIAL: NCT01413178
Title: A Randomized Trial to Compare Busulfan + Melphalan 140 mg/m2 With Melphalan 200 mg/m2 as Preparative Regimen for Autologous Hematopoietic Stem Cell Transplantation for Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0071; NCI-2011-02760 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Myeloma
Keywords: Myeloma; Multiple Myeloma; Light chain Multiple Myeloma; MM; Autologous Hematopoietic Stem Cell Transplantation; Busulfan; Busulfex; Myleran; Melphalan; Alkeran; G-CSF; Filgrastim; NeupogenTM; Questionnaire; Survey; Quality of Life; QOL
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Busulfan; Melphalan; Surveys and Questionnaires; Granulocyte Colony-Stimulating Factor; Filgrastim; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Busulfan + Melphalan (Experimental): Busulfan test dose (32 mg/m^2) on day -9 then 130 mg/m^2 intravenous (IV) Days -7, -6, -5, and -4 + Melphalan 70 mg/m2 IV on Days -2 and -1. Stem Cell Transplant (SCT) Day 0.
  Interventions: Drug: Busulfan; Drug: Melphalan; Other: Questionnaire; Drug: G-CSF; Procedure: Stem cell transplant
- Melphalan (Experimental): High-dose Melphalan 200 mg/m2/day IV over 30 minutes on day -2. SCT Day 0.
  Interventions: Other: Questionnaire; Drug: G-CSF; Drug: High Dose Melphalan; Procedure: Stem cell transplant

INTERVENTIONS:
Drug: Busulfan — Test dose (32 mg/m^2) on day -9 then 130 mg/m^2 by vein or adjusted dose on Days -7, -6, -5, and -4.
  Other Names: Busulfex; Myleran
  Arms: Busulfan + Melphalan
Drug: Melphalan — 70 mg/m2 by vein over 30 minutes minutes on Days -2 and -1.
  Other Names: Alkeran
  Arms: Busulfan + Melphalan
Other: Questionnaire — Quality of Life (QOL) questionnaire before starting the study drugs and then once every 4 weeks after the stem cell transplant, taking about 15 minutes to complete.
  Other Names: Survey
Drug: G-CSF — Approximately 5 mcg/kg/day subcutaneously beginning on Day +5.
  Other Names: Filgrastim; NeupogenTM
Drug: High Dose Melphalan — 200 mg/m2 by vein over 30 minutes on Day -2.
  Other Names: Alkeran
  Arms: Melphalan
Procedure: Stem cell transplant — Stem cell infusion on Day 0.
  Other Names: ABMT; autologous bone marrow transplantation; Peripheral Blood Progenitor Cells; PBPCs

SUMMARY:
The goal of this clinical research study is to compare Busulfex (busulfan) with or without Alkeran (melphalan) to learn which study therapy may be better at helping to control MM in patients who will receive an autologous stem cell transplant. The safety of this combination therapy will also be studied.

Melphalan and busulfan are designed to damage the DNA (genetic material) of cells, which may cause cancer cells to die.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups.

* Group 1 will receive melphalan and busulfan.
* Group 2 will receive melphalan.

Both groups will have a stem cell transplant.

Study Drug Administration:

If you are in Group 1, you will first receive an additional low-level "test" dose of busulfan given by vein to check how your blood levels change over time. This information will be used to decide the next dose that is needed to reach a target blood level of busulfan. Blood (about 1 teaspoon each time) will be drawn up to 11 times during the next 11 hours after the test dose and the first high-dose busulfan treatment.

A heparin lock line will be placed in a vein to lower the number of needle sticks needed for these draws.

This test dose of busulfan can be given as an outpatient before you are admitted to the hospital, or you will be admitted on Day -10 (10 days before your transplant) and will receive the test dose on Day -9. If it is not possible for these blood level tests to be performed for technical or scheduling reasons, you will receive the standard, fixed (unchanging) dose of busulfan.

Eight (8) or 10 days before the transplant, you will be admitted to the hospital and given hydration fluids by vein.

On Days -7, -6, -5, and -4, you will receive busulfan by vein over 3 hours. You will receive melphalan on Days -2 and -1 by vein over 30 minutes. You will receive the stem cell transplant through the CVC on Day 0.

If you are in Group 2, you may be admitted to the hospital 3 days before the transplant. You will receive hydration fluids by vein. Two (2) days before the transplant, you will receive melphalan by vein over 30 minutes. You will not receive melphalan the day before the transplant.

Stem Cell Transplant:

The day that you receive the stem cell transplant is called Day 0. The stem cells will be given by vein through the CVC. The cells will travel to your bone marrow where they are designed to start making healthy, new blood cells after several weeks. You will sign a separate consent for the collection of your stem cells.

Beginning 5 days after the transplant, you will receive filgrastim (G-CSF) through a needle under your skin 1 time each day until your blood cell levels return to normal. Filgrastim is designed to help with the growth of white blood cells.

You will be in the hospital after the transplant for about 2-4 weeks.

Questionnaire:

You will be asked to complete a quality-of-life questionnaire before starting the study drugs and then once a week during Weeks 1, 2, and 4 after the stem cell transplant. The questionnaire will take about 15 minutes to complete.

Follow-Up Visits:

About 3 months after the transplant, you will have a bone marrow aspiration and biopsy to check the status of the disease. To collect a bone marrow aspiration and biopsy, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.

Every 3 months during the first year after the transplant, blood (about 1-2 tablespoons) will be drawn to check your immune response and status of the disease.

About 1 year after the transplant, you will have a bone scan if the doctor thinks it is needed.

Length of Study:

One (1) year after the transplant, your participation in this study will be over.

If intolerable side effects from the chemotherapy occur or there is sign of disease after the transplant, you will be taken off study. If you have intolerable side effects after you receive chemotherapy, then you will still have the transplant. If you are taken off study early, you still may need to return for routine post-transplant follow-up visits, if your transplant doctor decides it is needed.

This is an investigational study. Busulfan and melphalan are commercially available and FDA approved for the treatment of myeloma. The use of melphalan alone before an autologous stem cell transplant is considered standard of care. Using busulfan with melphalan is investigational.

Up to 205 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple myeloma in complete remission (CR), partial remission (PR), or very good partial remission (VGPR), or symptomatic stable disease (no evidence of progression) including patients with light chain MM detected in the serum by free light chain assay.
2. Patients with non-secretory multiple myeloma [absence of a monoclonal protein (M protein) in serum as measured by electrophoresis (SPEP) and immunofixation (SIFE) and the absence of Bence Jones protein in the urine (UPEP) defined by use of conventional electrophoresis and immunofixation (UIFE) techniques] but with measurable disease on imaging studies like MRI, CT scan or PET scan.
3. Who have received at least two cycles of initial systemic therapy and are within 2 to 12 months of the first dose. Mobilization therapy is not considered initial therapy.
4. 70 years of age or younger.
5. Karnofsky performance score 70% or higher.
6. Cardiac function: left ventricular ejection fraction at rest > 40% within 3 months of registration.
7. Hepatic function: bilirubin < 2x the upper limit of normal and ALT and AST < 2.5x the upper limit of normal.
8. Renal function: creatinine clearance of >/= 40 mL/min, estimated or calculated.
9. Pulmonary function: DLCO, FEV1, FVC >/= 50% of predicted value (corrected for hemoglobin) within 3 months of registration
10. Signed informed consent form.

Exclusion Criteria:

1. Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and progression of clinical symptoms).
2. Patients seropositive for the human immunodeficiency virus (HIV).
3. Patients with history of myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
4. Patients participating in an investigational new drug protocol within 14 days before enrollment.
5. Female patients who are pregnant (positive b-HCG) or breastfeeding.
6. Prior stem cell transplantation allogeneic or autologous.
7. Prior organ transplant requiring immunosuppressive therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar H. Qazilbash, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bashir Q, Thall PF, Milton DR, Fox PS, Kawedia JD, Kebriaei P, Shah N, Patel K, Andersson BS, Nieto YL, Valdez BC, Parmar S, Rondon G, Delgado R, Hosing C, Popat UR, Oran B, Ciurea SO, Lin P, Weber DM, Thomas SK, Lee HC, Manasanch EE, Orlowski RZ, Williams LA, Champlin RE, Qazilbash MH. Conditioning with busulfan plus melphalan versus melphalan alone before autologous haemopoietic cell transplantation for multiple myeloma: an open-label, randomised, phase 3 trial. Lancet Haematol. 2019 May;6(5):e266-e275. doi: 10.1016/S2352-3026(19)30023-7. Epub 2019 Mar 22. PMID 30910541
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered in MD Anderson Cancer.
Groups:
- Busulfan + Melphalan: Busulfan with a target daily area under the curve (AUC) of 5000 with Melphalan 70 mg/m2 followed by a stem cell transplant
- Melphalan: High-dose Melphalan 200 mg/m2/day followed by a stem cell transplant
Period: Overall Study
Arm/Group | Busulfan + Melphalan | Melphalan
Started | 105 | 100
Completed | 104 | 98
Not Completed | 1 | 2
Not completed — Toxicity | 1 | 0
Not completed — Ineligible | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Busulfan + Melphalan | Melphalan | Total
Number analyzed (Participants) | 104 | 98 | 202
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58.9 [53.3 to 65.0] | 59.5 [51.9 to 64.2] | 59.2 [51.9 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 61 | 55 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 24 | 39
  White | 75 | 67 | 142
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 104 | 98 | 202

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Participants that are still alive and without Multiple Myeloma 3 years after Stem cell Transplantation.
Time Frame: 3 years after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Busulfan + Melphalan | Melphalan
Number analyzed (Participants) | 104 | 98
Participants | 72 | 50

2. Secondary Outcome: Number of Participants With Complete Response (CR)
Description: Complete response (CR), evaluated 90 days from transplant, defined as (i) negative immunofixation of the multiple myeloma (MM) protein in urine and serum, (ii) disappearance of any soft tissue plasmacytomas, and (iii) less than 5% plasma MM cells in the bone marrow. International Myeloma Working Group uniform response criteria.
Time Frame: Evaluated 90 days from transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Busulfan + Melphalan | Melphalan
Number analyzed (Participants) | 104 | 98
Participants | 12 | 15

3. Secondary Outcome: Treatment-Related Mortality (TRM) Between 2 Arms.
Time Frame: 100 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Busulfan + Melphalan | Melphalan
Number analyzed (Participants) | 104 | 98
Participants | 0 | 0

4. Secondary Outcome: Number of Participants That Had Grade 3-4 Toxicities.
Time Frame: At day 90 post SCT (Stem Cell Transplantation)
Measure: Number; unit: participants
Arm/Group | Busulfan + Melphalan | Melphalan
Number analyzed (Participants) | 104 | 98
participants
  Grade 3 - Diarrhea | 5 | 4
  Grade 3 - Elevated ALT | 3 | 0
  Grade 3 - Elevated Tbili | 2 | 0
  Grade 3 - Infection | 16 | 5
  Grade 3 - Mucositis | 15 | 0
  Grade 3 - Nausea | 5 | 2
  Grade 3 - Neuropathy | 1 | 0
  Grade 3 - Neutropenic fever | 73 | 32
  Grade 3 - Pneumonia | 1 | 1
  Grade 3 - Tachycardia | 1 | 0
  Grade 3 - Transient blindness | 1 | 0
  Grade 3 - Anorexia | 1 | 0
  Grade 3 - Myocardial ischemia | 1 | 1
  Grade 3 - Pleural effusion | 0 | 1
  Grade 3 - Rash | 0 | 1

5. Secondary Outcome: Overall Survival (OS)
Time Frame: From time of ASCT to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Busulfan + Melphalan | Melphalan
Number analyzed (Participants) | 104 | 98
Participants | 91 | 79

ADVERSE EVENTS:
Time Frame: From the time of ASCT until 12 months.
Arm/Group | Busulfan + Melphalan | Melphalan
All-Cause Mortality (participants affected / at risk) | 23/104 | 21/98
Serious Adverse Events (participants affected / at risk) | 73/104 | 32/98
Other Adverse Events (participants affected / at risk) | 101/104 | 98/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Busulfan + Melphalan (N=104) | Melphalan (N=98)
Diarrhea (Gastrointestinal disorders) | 5 | 4
Elevated ALT (Hepatobiliary disorders) | 3 | 0
Elevated Tbili (Hepatobiliary disorders) | 2 | 0
Infection (Infections and infestations) | 16 | 6
Mucositis (Gastrointestinal disorders) | 15 | 0
Myocardial ischemia (Cardiac disorders) | 1 | 1
Neuropathy (Nervous system disorders) | 1 | 0
Neutropenic fever (Infections and infestations) | 73 | 32
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Transient blindness (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Busulfan + Melphalan (N=104) | Melphalan (N=98)
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Chemo burns (Skin and subcutaneous tissue disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 57 | 82
Dizziness (Nervous system disorders) | 1 | 0
Dysuria (Reproductive system and breast disorders) | 1 | 0
Elevated ALT (Hepatobiliary disorders) | 31 | 1
Elevated AST (Hepatobiliary disorders) | 1 | 1
Elevated creatinine (Blood and lymphatic system disorders) | 3 | 0
Elevated Tbili (Hepatobiliary disorders) | 8 | 9
Fever (Infections and infestations) | 17 | 8
Fluid overload (Cardiac disorders) | 63 | 22
Headache (Nervous system disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 3 | 2
Hypertension (Cardiac disorders) | 16 | 5
Hypotension (Cardiac disorders) | 1 | 0
Infection (Infections and infestations) | 18 | 17
Mucositis (Gastrointestinal disorders) | 86 | 49
Nausea (Gastrointestinal disorders) | 99 | 98
Neutropenic fever (Infections and infestations) | 1 | 33
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 4
Tachycardia (Cardiac disorders) | 4 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Weakness of extremities (Musculoskeletal and connective tissue disorders) | 1 | 0
Anorexia (Psychiatric disorders) | 0 | 3
involuntary leg movements (Musculoskeletal and connective tissue disorders) | 0 | 1
Lip ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Myocardial ischemia (Cardiac disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT01413178/Prot_SAP_000.pdf